CLINICAL TRIAL: NCT01445808
Title: Psychodynamic Motivation and Training Program (PMT) as Secondary Prevention in Patients With Stable Coronary Heart Disease
Brief Title: Psychodynamic Motivation and Training Program
Acronym: PMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Matthias Michal, PD Dr. med., Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB 837.274.11 (7816)
Record Dates: First submitted 2011-09-30; First posted 2011-10-04 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Coronary Heart Disease; Physical Activity
Keywords: psychodynamic psychotherapy; coronary heart disease; physical activity; secondary prevention
MeSH Terms: conditions — Coronary Disease; Motor Activity | interventions — Counseling; Exercise; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Psychodynamic Motivation and Training Program (PMT) (Experimental)
  Interventions: Behavioral: Psychodynamic Motivation and Training Program (PMT)
- Advice in Exercise Training (Active Comparator): One session of advice in exercise training based on the results of spiroergometry
  Interventions: Behavioral: Advice in Exercise Training (+Ex)
- Treatment as usual (TAU) (Other): Usual care by family doctor and cardiologist
  Interventions: Other: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Psychodynamic Motivation and Training Program (PMT) — The Psychodynamic Motivation and Training Program (PMT) is a psychodynamic stepped care approach. Depending on the individual needs PMT consists of 3 to 8 sessions of individual psychodynamic psychotherapy. If appropriate session 4 - 8 may be conducted by a nurse. PMT targets the mental and external barriers to improve physical activity by focusing on affects, interpersonal relations and maladaptive self- and other representations. PMT will be offered in addition to +Ex.
  Arms: Psychodynamic Motivation and Training Program (PMT)
Behavioral: Advice in Exercise Training (+Ex) — Advice in Exercise Training consists of one individual session of advice in exercise training based on the results of the spiroergometry.
  Arms: Advice in Exercise Training
Other: Treatment as usual (TAU) — Usual care by family doctor, cardiologist
  Arms: Treatment as usual (TAU)

SUMMARY:
The purpose of this study is to examine the effectiveness of a Psychodynamic Motivation and Training Program (PMT) for the improvement of physical fitness in patients with stable coronary heart disease as compared to advice in exercise training or treatment as usual.

DETAILED DESCRIPTION:
Nonpharmacological secondary prevention of coronary heart disease is considered to be a safe and effective measure for reducing mortality substantially. Major targets are the improvement of physical activity and dietary habits, smoking cessation and stress reduction. Despite the effectiveness of life style changes, the compliance rate of patients is very low. To improve compliance with life style change programs psychotherapeutic interventions appear to have significant potential. Against this background our study aims to examine the effectiveness of a Psychodynamic Motivation and Training Program (PMT) in addition to one session of advice in exercise training based on the results of spiroergometry (+EX) and usual cardiological care (TAU). PMT will be compared with +Ex and TAU. N = 90 patients with stable coronary artery disease class, low physical activity, class I to III angina pectoris will be randomly assigned to the three treatment conditions. The Primary efficacy endpoint is change in the anaerobic threshold from baseline to 6 month follow-up. The results of the study will 1) help to determine the effectiveness of a psychodynamic life style change programs for the secondary prevention of cardiovascular disease and 2) will help to identify measures for designing specifically tailored interventions to improve compliance with cardiovascular prevention.

ELIGIBILITY:
Inclusion Criteria:

* Stable coronary heart disease with CCS functional classification of angina class I-III
* Low self rated physical activity
* Condition after percutaneous coronary intervention > 4 weeks until < 26 weeks or > 52 weeks after index percutaneous coronary intervention
* Residence < 50 km radius of Mainz
* If treatment with betablockers or ivabradine then stable > 4 weeks

Exclusion Criteria:

* Acute coronary sydnrome or myocardial infarction < 8 weeks
* Coronary stenosis of the dominant vessel > 25% or high grade stenosis of the left coronary artery
* Heart failure with left ventricular ejection fraction < 40%
* NYHA III-IV
* Severe heart valve disorder
* Insulin dependent diabetes
* Orthopedic disorders or other disorders, which preclude regular physical activity
* Coronary artery bypass surgery < 6 months before index PCI
* Severe obesity (BMI ≥ 40)
* Need for systemic immunosuppression with cortisone or methotrexate
* Kidney failure with need for dialysis
* Intake of nitrates < 12 hours

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-10; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change in individual anaerobic threshold according to lactate kinetics during spiroergometry | 6 months

SECONDARY OUTCOMES:
Change in quality of life according to the EQ-5D | 6 months
Change in the severity of impairment by angina symptoms according to the Seattle Angina Questionnaire | 6 Months
Change in the self-rated habitual physical activity according to the Habitual Physical Activity Questionnaire | 6 months
Change in endothelial function according to the flow mediated dilatation | 6 months
Change in high density lipoprotein levels | 6 months
Change in biomarkers of inflammation and oxidative burst | 6 months
Change in fatigue according to the Maastricht Questionnaire | 6 months
Change in illness perception | 6 months
  (Illness perception as measured with the Brief Illness Perception Questionnaire)
Change in maximal aerobic capacity (VO2 max) | 6 months
Change in body mass index | 6 months
  (BMI kg/m²)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Michal, PD Dr. med., Principal Investigator — University Medical Center Mainz, Department of Psychosomatic Medicine and Psychotherapy
Locations (1):
- University Medical Center Mainz, Mainz, Germany

REFERENCES:
- [Derived] Michal M, Simon P, Gori T, Konig J, Wild PS, Wiltink J, Tug S, Sterzing B, Unterrainer J, Munzel T, Beutel ME. Psychodynamic Motivation and Training program (PMT) for the secondary prevention in patients with stable coronary heart disease: study protocol for a randomized controlled trial of feasibility and effects. Trials. 2013 Sep 25;14:314. doi: 10.1186/1745-6215-14-314. PMID 24066805